CLINICAL TRIAL: NCT05804552
Title: The Effect of Dorsal Genital Nerve Stimulation on Opening Urethral Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thea Christoffersen (Other)
Collaborators: InnoCon Medical (Industry)
Responsible Party: Sponsor-Investigator, Thea Christoffersen, Medical Doctor, Principal Investigator, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-22063824
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Stress Urinary Incontinence
Keywords: Electrical Stimulation; Urethral pressure; Neuromodulation
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dorsal genital nerve stimulation (Experimental)
  Interventions: Device: Dorsal genital nerve stimulation

INTERVENTIONS:
Device: Dorsal genital nerve stimulation — Two types of stimulation electrodes will be used: UCon Patch Electrodes (InnoCon Medical ApS, Denmark) and ValuTrodes/EconoStim Electrodes (5x5 cm, Axelgaard Manufacturing Co. Ltd., United States). The UCon Patch Electrode acts as a cathode and will be placed on the clitoris. The ValuTrode/EconoStim acts as an anode and will be placed on the lower abdomen. The continuous stimulation consists of a train of single pulses provided continuously with a frequency of 20 Hz and a pulse duration of 200 μs. The burst stimulus pattern consists of a train of bursts. The length of the train is 10 s and will consist of 20-30 bursts/s. One burst consists of 5 identical square pulses (monophasic). The inter-pulse interval is 4 ms (time between the onset of 2 consecutive pulses) while a pulse duration of 200 μs will be used.

SUMMARY:
This study aims to investigate the effect of electrical stimulation of the dorsal genital nerve on the urethral pressure in healthy women.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight (Body weight 50 kg or more, Body Mass Index 18-5-30 kg/m2)
* Signed an informed consent

Exclusion Criteria:

Any history of clinically significant diseases, unless regarded irrelevant and/or stable by the investigator

* Any history or evidence of clinically significant urinary incontinence, urinary retention, overactive bladder, or other voiding dysfunction
* Known or suspected nerve injuries or paraesthesia in the pelvic area
* Pregnancy within six months before enrolment
* Breastfeeding within three months before enrolment
* Smoking or other regular use of any form of nicotine product during the study period and the previous 3 months
* Current or prior participation (within 3 months before screening) in other clinical trials that might affect the results of this study (judged by the investigator)
* Any systemic drug use within 2 weeks before the first study day (prescription drugs, over-the-counter drugs, herbal drugs, and/or illicit drugs), except for occasional use of paracetamol (up to 4 g/day), ibuprofen, or antihistamine, hormonal contraceptives and hormone replacement therapy.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender identidy
Enrollment: 10 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Effect of burst dorsal genital nerve stimulation compared to baseline | Baseline and during dorsal genital nerve stimulation
  The difference in mean opening urethral pressure (in cmH20) measured with urethral pressure reflectometry during electrical burst stimulation of dorsal genital nerve (reflex-induced pelvic floor contraction) compared to mean baseline opening urethral pressure during squeezing condition

SECONDARY OUTCOMES:
Effect of continuous dorsal genital nerve stimulation on resting pressure compared to baseline | Baseline and during dorsal genital nerve stimulation
  The difference in mean opening urethral pressure (in cmH20) measured with urethral pressure reflectometry during maximal tolerated continuous dorsal genital nerve stimulation compared to mean baseline OUP (resting condition).
Effect of continuous dorsal genital nerve stimulation on squeezing pressure compared to baseline | Baseline and during dorsal genital nerve stimulation
  The difference in mean opening urethral pressure (in cmH20) measured with urethral pressure reflectometry during maximal tolerated continuous dorsal genital nerve stimulation compared to mean baseline opening urethral pressure (squeezing condition).

CONTACTS AND LOCATIONS:
Locations (1):
- Zelo Phase 1 unit, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No